CLINICAL TRIAL: NCT02122770
Title: A Phase 1 Study to Evaluate the Effects of Fluconazole and Itraconazole CYP3A-Mediated Inhibition on the Pharmacokinetics, Safety, and Tolerability of MLN4924 in Patients With Advanced Solid Tumors
Brief Title: Effects of Fluconazole and Itraconazole CYP3A-Mediated Inhibition on the Pharmacokinetics, Safety, and Tolerability of MLN4924 in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C15011; U1111-1155-6191 (Other: World Health Organization)
Record Dates: First submitted 2014-04-23; First posted 2014-04-25 (Estimated); Results first posted 2019-01-07 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2018-06

CONDITIONS: Advanced Solid Tumors
Keywords: Drug Therapy
MeSH Terms: interventions — pevonedistat; Fluconazole; Itraconazole; Docetaxel; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MLN4924 + Fluconazole (Experimental): Part A: MLN4924, 8 milligram per square meter (mg/m^2), intravenously, once on Days 1 and 8; and fluconazole, 400 milligram (mg), tablets, orally, once on Day 4, and 200 mg, once daily on Days 5-10.
  Part B: MLN4924, at a dose previously deemed tolerable, given on Days 1, 3, and 5 of each 21-day Cycle (Study C15010, Clinicaltrials.gov Identifier # NCT01862328) in combination with docetaxel or carboplatin + paclitaxel at standard dose regimen on Day 1 of each 21-day Cycle.
  Interventions: Drug: MLN4924; Drug: Fluconazole; Drug: Docetaxel; Drug: Carboplatin; Drug: Paclitaxel
- MLN4924 + Itraconazole (Experimental): Part A: MLN4924, 8-mg/m^2, intravenously, once on Days 1 and 8; and itraconazole, 200 mg, oral solution, once daily on Days 4-10.
  Part A (safety lead-in step): MLN4924, 15mg/m^2, intravenously, once on Days 1 and 8; and itraconazole, 200 mg, oral solution, once daily on Days 4-10.
  Part A: MLN4924, 20mg/m^2, intravenously, once on Days 1 and 8; and itraconazole, 200 mg, oral solution, once daily on Days 4-10.
  Part B: MLN4924, at a dose previously deemed tolerable given, on Days 1, 3, and 5 of each 21-day Cycle (Study C15010, ClinicalTrails.gov Identifier # NCT01862328) in combination with docetaxel or carboplatin + paclitaxel at standard dose regimen on Day 1 of each 21-day Cycle.
  Interventions: Drug: MLN4924; Drug: Itraconazole; Drug: Docetaxel; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: MLN4924 — MLN4924 intravenous solution.
Drug: Fluconazole — Fluconazole tablets.
  Arms: MLN4924 + Fluconazole
Drug: Itraconazole — Itraconazole oral solution.
  Arms: MLN4924 + Itraconazole
Drug: Docetaxel — Docetaxel intravenous solution.
Drug: Carboplatin — Carboplatin intravenous solution.
Drug: Paclitaxel — Paclitaxel intravenous solution.

SUMMARY:
The primary purpose of this study is to assess the effect of multiple-dose administration of fluconazole on the single-dose intravenous (IV) pharmacokinetics (PK) of MLN4924; and to assess the effect of multiple-dose administration of itraconazole on the single-dose IV PK of MLN4924.

DETAILED DESCRIPTION:
The drug being tested in this study is MLN4924. MLN4924 is being evaluated to assess drug-drug interactions (DDIs) with the moderate and strong CYP3A inhibitors, fluconazole and itraconazole, respectively, in participants with advanced solid tumors. This study will look at the blood concentrations of MLN4924 as it relates to treatment with fluconazole and itraconazole.

The study will enroll approximately 52 participants. In Part A, participants will be administered MLN4924 via a 1-hour (+- 5 minutes) intravenous (IV) infusion in combination with either fluconazole or itraconazole administered orally. After participants complete Part A, they will have the opportunity to begin treatment in Part B. In Part B, participants will be administered MLN4924 via a 1-hour (+- 5 minutes) IV infusion in combination with either docetaxel or carboplatin + paclitaxel, the three of which would also be administered intravenously.

This multi-center trial will be conducted in the United States. Participation in Part A of this study will include a screening visit and two weeks of treatment; participation in Part B of this study will include up to an 8-week drug washout period (from last dosing in Part A) and treatment until participants experience symptomatic deterioration, progressive disease, until treatment is discontinued for another reason, or until the study is stopped.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants 18 years of age or older.
2. Must have a histologically or cytologically confirmed metastatic or locally advanced and incurable solid tumor that is deemed appropriate for treatment with 1 of the 2 chemotherapy regimens in Part B of this study, or have progressed despite standard therapy, or for whom conventional therapy is not considered effective. The tumor must be radiographically or clinically evaluable or measurable.
3. Recovered (that is, less than or equal to (<=) Grade 1 toxicity) from the effects of prior antineoplastic therapy.
4. Suitable venous access for the study-required blood sampling for MLN4924 pharmacokinetic (PK) and pharmacodynamic assessments.
5. Eastern Cooperative Oncology Group performance status (PS) of 0 or 1.
6. Clinical laboratory values as specified below within 3 days before the first dose of study drug:

   1. Hemoglobin greater than or equal to (>=) 9 gram per deciliter (g/dL)
   2. Absolute neutrophil count >=1,500 per cubic millimeter (/mm^3), not supported by growth factor
   3. Platelet count >=100,000/mm^3
   4. Total bilirubin <=upper limit of normal (ULN)
   5. Prothrombin time (PT) and activated partial thromboplastin time (aPTT) <=1.5*ULN
   6. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) <=2.5*ULN

      • For participants to be treated with MLN4924 + docetaxel in Part B, AST and ALT must be <=1.5*ULN, and total bilirubin should be within the normal range.
   7. Serum creatinine <=1.2 mg/dL or calculated/measured creatinine clearance >=50 mL/minute
7. Female participants who:

   1. Are postmenopausal for at least 1 year before the screening visit, OR
   2. Are surgically sterile, OR
   3. If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through four months after the last dose of study drug, or
   4. Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [example, calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)
   5. Male participants, even if surgically sterilized (that is, status postvasectomy), who:
   6. Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug, or
   7. Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [example, calendar, ovulation, symptothermal, postovulation methods for the female partner] and withdrawal are not acceptable methods of contraception.)
8. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.
9. Participants who are willing to refrain from donating blood for at least 90 days after their final dose of MLN4924 and (for male participants) willing to refrain from donating semen for at least 4 months after their final dose of MLN4924.

Exclusion Criteria:

1. Prior treatment with MLN4924; however, prior treatment with docetaxel, paclitaxel, and carboplatin is allowed.
2. Treatment with any systemic antineoplastic therapy or investigational products within 21 days before the first dose of study treatment.
3. Radiotherapy within 14 days before the first dose of study treatment.
4. Prior treatment with radiation therapy involving >= 25 percent (%) of hematopoietically active bone marrow.
5. Known hypersensitivity or history of severe intolerance or toxicity to study-assigned chemotherapy. Note: History of severe hypersensitivity reactions to docetaxel (polysorbate 80-based formulations) for participants to be treated with MLN4924 + docetaxel; history of hypersensitivity to carboplatin for participants to be treated with MLN4924 + carboplatin + paclitaxel; or history of severe hypersensitivity to paclitaxel (Cremophor-based formulations) for participants to be treated with MLN4924 + carboplatin + paclitaxel in Part B.
6. Known hypersensitivity/allergy to fluconazole or itraconazole or their respective excipients.
7. Systemic treatment with moderate and strong cytochrome P450 (CYP) CYP3A inhibitors or inducers must be discontinued at least 14 days before the first dose of MLN4924. Moderate and strong CYP3A inhibitors and CYP3A inducers are not permitted during the study. Participants must have no history of amiodarone use in the 6 months before the first dose of MLN4924.
8. Any life-threatening or serious medical or psychiatric illness unrelated to cancer that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
9. Major surgery within 14 days before the first dose of study treatment.
10. Active uncontrolled infection or severe infectious disease, such as pneumonia, meningitis, septicemia, or methicillin-resistant Staphylococcus aureus infection.
11. Clinically significant central nervous system disease defined as untreated, progressive, or requiring steroids for control of symptoms.
12. Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of fluconazole or itraconazole including difficulty swallowing capsules.
13. Persistent diarrhea (>= Grade 2) lasting greater than (>) 3 days within 2 weeks before the first dose of study treatment.
14. Known hepatic cirrhosis, hepatitis B surface antigen-positive status, or suspected active hepatitis C infection. Note: Participants who have isolated positive hepatitis B core antibody (that is, in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody) must have an undetectable hepatitis B viral load.
15. Known human immunodeficiency virus (HIV) positive status.
16. Female participants who are lactating and breastfeeding or have a positive serum pregnancy test during the Screening period or a positive urine pregnancy test on Day 1 before first dose of study drug.
17. Uncontrolled high blood pressure (that is, systolic blood pressure >180 millimeter of mercury [mmHg], diastolic blood pressure >95 mmHg).
18. Left ventricular ejection fraction < 50% as assessed by echocardiogram or radionuclide angiography.
19. Congestive heart failure New York Heart Association Class III or IV, or Class II with a recent decompensation requiring hospitalization within 4 weeks before screening.
20. Cardiomyopathy or history of ischemic heart disease.

    o Participants with ischemic heart disease who have had acute coronary syndrome (ACS), myocardial infarction (MI), or revascularization (example, coronary artery bypass graft, stent) in the past 6 months are excluded. However, participants with ischemic heart disease who have had ACS, MI, or revascularization greater than 6 months before screening and who are without cardiac symptoms may enroll.
21. Arrhythmia (example, history of polymorphic ventricular fibrillation or torsade de pointes). However, participants with < Grade 3 atrial fibrillation for a period of at least 6 months may enroll. Grade 3 atrial fibrillation is defined as symptomatic and incompletely controlled medically, or controlled with device (example, pacemaker) or ablation, and is excluded. Participants with paroxysmal atrial fibrillation are permitted to enroll.
22. Prolonged rate corrected QT interval (QTc) >=500 millisecond (msec), calculated according to institutional guidelines.
23. Implantable cardioverter defibrillator.
24. Participants with a cardiac pacer whose heart rate is set at a fixed rate and participants on concomitant medication that may limit increase in heart rate in response to hypotension (example, high-dose beta blocker).
25. Moderate to severe aortic or mitral stenosis or other valvulopathy (ongoing).
26. Known moderate to severe chronic obstructive pulmonary disease (COPD), interstitial lung disease, pulmonary fibrosis, and pulmonary arterial hypotension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2017-06-05 (Actual); Study Completion 2017-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Millennium Pharmaceuticals, Inc.
Locations (4):
- United States (4):
  - Winship Cancer Institute at Emory University, Atlanta, Georgia
  - Siteman Cancer Center - South County, St Louis, Missouri
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Mary Crowley Medical Research Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 investigative site in the United States from 01 April 2014 to 05 June 2017.
Pre-assignment Details: Participants with advanced solid tumors were enrolled in this study to receive MLN4924. This study included 2 parts: Part A (drug-drug interaction)- participants received MLN4924 with fluconazole or itraconazole and in Part B (standard of care)- participants received MLN4924 in combination with docetaxel or carboplatin and paclitaxel.
Groups:
- Part A: MLN4924 8 mg/m^2 + Fluconazole 400 mg: MLN4924 8 milligram per square meter (mg/m^2), infusion, intravenously, once on Days 1 and 8 along with fluconazole, 400 milligram (mg), tablets, orally, once on Day 4, and 200 mg, once daily on Days 5-10.
- Part A: MLN4924 8 mg/m^2 + Itraconazole 200 mg: MLN4924 8 mg/m^2, infusion, intravenously, once on Days 1 and 8 along with itraconazole, 200 mg, solution, orally, once daily on Days 4-10.
- Part A: MLN4924 15 mg/m^2 + Itraconazole 200 mg: MLN4924 15 mg/m^2, infusion, intravenously, once on Days 1 and 8 along with itraconazole, 200 mg, solution, orally, once daily on Days 4-10.
- Part A: MLN4924 20 mg/m^2 + Itraconazole 200 mg: MLN4924 20 mg/m^2, infusion, intravenously, once on Days 1 and 8 along with itraconazole, 200 mg, solution, orally, once daily on Days 4-10.
- Part B: MLN4924 + Docetaxel: MLN4924, 8-20 mg/m^2, on Days 1, 3, and 5 along with docetaxel at standard dose regimen on Day 1 of a 21-day treatment Cycle until symptomatic deterioration, progressive disease (PD), treatment discontinuation, or until the study is stopped.
- Part B: MLN4924 + Carboplatin or Paclitaxel: MLN4924, 8-20 mg/m^2, on Days 1, 3, and 5 along with carboplatin or paclitaxel at standard dose regimen on Day 1 of a 21-day treatment Cycle until symptomatic deterioration, progressive disease (PD), treatment discontinuation, or until the study is stopped.
Period: Part A: Drug-drug Interaction 2
Arm/Group | Part A: MLN4924 8 mg/m^2 + Fluconazole 400 mg | Part A: MLN4924 8 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 15 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 20 mg/m^2 + Itraconazole 200 mg | Part B: MLN4924 + Docetaxel | Part B: MLN4924 + Carboplatin or Paclitaxel
Started | 13 | 13 | 6 | 19 | 0 | 0
Completed (Completed Part A, ongoing to Part B) | 9 | 7 | 4 | 16 | 0 | 0
Not Completed | 4 | 6 | 2 | 3 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 1 | 2 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Symptomatic Deterioration | 1 | 5 | 0 | 1 | 0 | 0
Period: Part B: Standard of Care
Arm/Group | Part A: MLN4924 8 mg/m^2 + Fluconazole 400 mg | Part A: MLN4924 8 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 15 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 20 mg/m^2 + Itraconazole 200 mg | Part B: MLN4924 + Docetaxel | Part B: MLN4924 + Carboplatin or Paclitaxel
Started | 0 | 0 | 0 | 0 | 23 | 13
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 23 | 13
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 4 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 4 | 2
Not completed — Symptomatic Deterioration | 0 | 0 | 0 | 0 | 5 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 10 | 8

BASELINE CHARACTERISTICS:
Population: The safety population for Part A included all enrolled participants who received at least 1 dose of MLN4924 during Part A.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: MLN4924 8 mg/m^2 + Fluconazole 400 mg | Part A: MLN4924 8 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 15 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 20 mg/m^2 + Itraconazole 200 mg | Total
Number analyzed (Participants) | 13 | 13 | 6 | 19 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 1 | 11 | 26
  >=65 years | 5 | 7 | 5 | 8 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 4 | 8 | 27
  Male | 6 | 5 | 2 | 11 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 10 | 6 | 14 | 43
  Unknown or Not Reported | 0 | 3 | 0 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 2 | 3 | 8
  White | 11 | 10 | 4 | 16 | 41
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 13 | 6 | 19 | 51
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 165.82 (12.142) | 166.49 (10.023) | 167.93 (6.998) | 171.46 (9.399) | 168.34 (10.122)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 71.22 (24.051) | 64.21 (16.536) | 76.58 (16.616) | 87.55 (32.311) | 76.15 (26.471)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: square meter (m^2)] | 1.792 (0.3405) | 1.712 (0.2384) | 1.883 (0.2297) | 2.021 (0.3736) | 1.868 (0.3372)

OUTCOME MEASURES:

1. Primary Outcome: Part A Cmax: Maximum Observed Plasma Concentration for MLN4924 and MLN4924 + Fluconazole
Time Frame: Day 1 (MLN4924) and Day 8 (MLN4924 + Fluconazole): pre-dose and at multiple time points (up to 72 hours) post-dose
Population: The pharmacokinetic (PK) evaluable population included all enrolled participants who received all protocol-specified dose regimens within each period during Part A, did not received any excluded medications throughout the completion of PK sampling, and had sufficient MLN4924 plasma concentration-time data to estimate PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Part A: MLN4924 8 mg/m^2: MLN4924 8 mg/m^2, infusion, intravenously, once on Day 1.
- Part A: MLN4924 8 mg/m^2 + Fluconazole 400 mg: MLN4924 8 mg/m^), infusion, intravenously, once on Day 8 along with fluconazole, 400 milligram (mg), tablets, orally, once on Day 4, and 200 mg, once daily on Days 5-10.
Arm/Group | Part A: MLN4924 8 mg/m^2 | Part A: MLN4924 8 mg/m^2 + Fluconazole 400 mg
Number analyzed (Participants) | 12 | 12
nanogram per milliliter (ng/mL) | 51.6 (52.3) | 51.0 (30.8)
Statistical Analysis 1: Comparison: Part A: MLN4924 8 mg/m^2 vs Part A: MLN4924 8 mg/m^2 + Fluconazole 400 mg; Natural-log transformed pharmacokinetic parameters were fit using a mixed effects model with study day as a fixed effect and participant as a random effect. Geometric least square (LS) means and geometric LS mean ratio were back-transformed least squares mean and treatment mean difference; Test type: Superiority; Geometric LS Mean Ratio = 98.75, 90% CI 2-sided [82.60 to 118.05]

2. Primary Outcome: Part A AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for MLN4924 and MLN4924 + Fluconazole
Time Frame: Day 1 (MLN4924) and Day 8 (MLN4924 + Fluconazole): pre-dose and at multiple time points (up to 72 hours) post-dose
Population: The PK evaluable population included all enrolled participants who received all protocol-specified dose regimens within each period during Part A, did not received any excluded medications throughout the completion of PK sampling, and had sufficient MLN4924 plasma concentration-time data to estimate PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Part A: MLN4924 8 mg/m^2 | Part A: MLN4924 8 mg/m^2 + Fluconazole 400 mg
Number analyzed (Participants) | 12 | 12
hour*nanogram per milliliter (h*ng/mL) | 445 (16.7) | 491 (15.5)
Statistical Analysis 1: Comparison: Part A: MLN4924 8 mg/m^2 vs Part A: MLN4924 8 mg/m^2 + Fluconazole 400 mg; Natural-log transformed pharmacokinetic parameters were fit using a mixed effects model with study day as a fixed effect and participant as a random effect. Geometric LS means and geometric LS mean ratio were back-transformed least squares mean and treatment mean difference; Test type: Superiority; Geometric LS Mean Ratio = 110.21, 90% CI 2-sided [102.34 to 118.69]

3. Primary Outcome: Part A AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for MLN4924 and MLN4924 + Fluconazole
Time Frame: Day 1 (MLN4924) and Day 8 (MLN4924 + Fluconazole): pre-dose and at multiple time points (up to 72 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A: MLN4924 8 mg/m^2 | Part A: MLN4924 8 mg/m^2 + Fluconazole 400 mg
Number analyzed (Participants) | 12 | 12
h*ng/mL | 450 (16.8) | 498 (15.9)
Statistical Analysis 1: Comparison: Part A: MLN4924 8 mg/m^2 vs Part A: MLN4924 8 mg/m^2 + Fluconazole 400 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Geometric LS Mean Ratio = 110.66, 90% CI 2-sided [102.53 to 119.43]

4. Primary Outcome: Part A Cmax: Maximum Observed Plasma Concentration for MLN4924 and MLN4924 + Itraconazole
Time Frame: Day 1 (MLN4924) and Day 8 (MLN4924 + Itraconazole): pre-dose and at multiple time points (up to 72 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part A: MLN4924 8 mg/m^2 + Itraconazole 200 mg: MLN4924 8 mg/m^2, infusion, intravenously, once on Day 8 along with itraconazole, 200 mg, solution, orally, once daily on Days 4-10.
- Part A: MLN4924 15 mg/m^2: MLN4924 15 mg/m^2, infusion, intravenously, once on Day 1.
- Part A: MLN4924 15 mg/m^2 + Itraconazole 200 mg: MLN4924 15 mg/m^2, infusion, intravenously, once on Day 8 along with itraconazole, 200 mg, solution, orally, once daily on Days 4-10.
- Part A: MLN4924 20 mg/m^2: MLN4924 20 mg/m^2, infusion, intravenously, once on Day 1.
- Part A: MLN4924 20 mg/m^2 + Itraconazole 200 mg: MLN4924 20 mg/m^2, infusion, intravenously, once on Day 8 along with itraconazole, 200 mg, solution, orally, once daily on Days 4-10.
Arm/Group | Part A: MLN4924 8 mg/m^2 | Part A: MLN4924 8 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 15 mg/m^2 | Part A: MLN4924 15 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 20 mg/m^2 | Part A: MLN4924 20 mg/m^2 + Itraconazole 200 mg
Number analyzed (Participants) | 13 | 13 | 6 | 6 | 14 | 14
ng/mL | 59.1 (52.4) | 66.8 (53.7) | 121 (61.0) | 193 (46.9) | 178 (76.3) | 137 (29.9)
Statistical Analysis 1: Comparison: Part A: MLN4924 8 mg/m^2 vs Part A: MLN4924 8 mg/m^2 + Itraconazole 200 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Geometric LS Mean Ratio = 113.05, 90% CI 2-sided [85.35 to 149.74]
Statistical Analysis 2: Comparison: Part A: MLN4924 15 mg/m^2 vs Part A: MLN4924 15 mg/m^2 + Itraconazole 200 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Geometric LS Mean Ratio = 159.55, 90% CI 2-sided [89.97 to 282.96]
Statistical Analysis 3: Comparison: Part A: MLN4924 20 mg/m^2 vs Part A: MLN4924 20 mg/m^2 + Itraconazole 200 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Geometric LS Mean Ratio = 77.26, 90% CI 2-sided [55.19 to 108.17]

5. Primary Outcome: Part A AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for MLN4924 and MLN4924 + Itraconazole
Time Frame: Day 1 (MLN4924) and Day 8 (MLN4924 + Itraconazole): pre-dose and at multiple time points (up to 72 hours) post-dose
Population: PK population:enrolled participants who received all protocol-specified dose regimens within each period in Part A,did not receive any excluded medications throughout completion of PK sampling, had sufficient MLN4924 plasma concentration-time data to estimate PK parameters. PK analysis population where data at specified time points were available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A: MLN4924 8 mg/m^2 | Part A: MLN4924 8 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 15 mg/m^2 | Part A: MLN4924 15 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 20 mg/m^2 | Part A: MLN4924 20 mg/m^2 + Itraconazole 200 mg
Number analyzed (Participants) | 13 | 13 | 6 | 6 | 14 | 14
h*ng/mL | 459 (24.7) | 571 (23.5) | 793 (18.2) | 1030 (17.3) | 1110 (30.2) | 1140 (22.7)
Statistical Analysis 1: Comparison: Part A: MLN4924 8 mg/m^2 vs Part A: MLN4924 8 mg/m^2 + Itraconazole 200 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Geometric LS Mean Ratio = 121.57, 90% CI 2-sided [110.92 to 133.24]
Statistical Analysis 2: Comparison: Part A: MLN4924 15 mg/m^2 vs Part A: MLN4924 15 mg/m^2 + Itraconazole 200 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Geometric LS Mean Ratio = 130.16, 90% CI 2-sided [106.99 to 158.35]
Statistical Analysis 3: Comparison: Part A: MLN4924 20 mg/m^2 vs Part A: MLN4924 20 mg/m^2 + Itraconazole 200 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Geometric LS Mean Ratio = 101.36, 90% CI 2-sided [90.72 to 113.23]

6. Primary Outcome: Part A AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for MLN4924 and MLN4924 + Itraconazole
Time Frame: Day 1 (MLN4924) and Day 8 (MLN4924 + Itraconazole): pre-dose and at multiple time points (up to 72 hours) post-dose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A: MLN4924 8 mg/m^2 | Part A: MLN4924 8 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 15 mg/m^2 | Part A: MLN4924 15 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 20 mg/m^2 | Part A: MLN4924 20 mg/m^2 + Itraconazole 200 mg
Number analyzed (Participants) | 13 | 13 | 6 | 6 | 14 | 14
h*ng/mL | 465 (25.1) | 585 (23.9) | 798 (18.1) | 1060 (16.1) | 1120 (30.4) | 1130 (23.5)
Statistical Analysis 1: Comparison: Part A: MLN4924 8 mg/m^2 vs Part A: MLN4924 8 mg/m^2 + Itraconazole 200 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Geometric LS Mean Ratio = 122.95, 90% CI 2-sided [112.13 to 134.82]
Statistical Analysis 2: Comparison: Part A: MLN4924 15 mg/m^2 vs Part A: MLN4924 15 mg/m^2 + Itraconazole 200 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Geometric LS Mean Ratio = 130.16, 90% CI 2-sided [106.99 to 158.35]
Statistical Analysis 3: Comparison: Part A: MLN4924 20 mg/m^2 vs Part A: MLN4924 20 mg/m^2 + Itraconazole 200 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Geometric LS Mean Ratio = 100.89, 90% CI 2-sided [91.14 to 111.68]

7. Secondary Outcome: Part A: Plasma Clearance (CLp) for MLN4924
Time Frame: Days 1 and 8: predose and at multiple time-points (up to 72 hours) postdose for Part A
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | Part A: MLN4924 8 mg/m^2 + Fluconazole 400 mg | Part A: MLN4924 8 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 15 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 20 mg/m^2 + Itraconazole 200 mg
Number analyzed (Participants) | 12 | 13 | 6 | 14
liter per hour (L/h)
  Day 1 | 31.7 (24.9) | 29.2 (27.5) | 35.2 (16.3) | 35.8 (41.6)
  Day 8: number analyzed (Participants) | 12 | 12 | 6 | 14
  Day 8 | 28.6 (30.2) | 23.2 (32.5) | 26.5 (18.6) | 35.5 (33.6)

8. Secondary Outcome: Part A Tmax: Time to Reach the Cmax for MLN4924
Time Frame: Days 1 and 8: predose and at multiple time-points (up to 72 hours) postdose for Part A
Population: as for outcome 5
Measure: Median (Full Range); unit: hour
Arm/Group | Part A: MLN4924 8 mg/m^2 + Fluconazole 400 mg | Part A: MLN4924 8 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 15 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 20 mg/m^2 + Itraconazole 200 mg
Number analyzed (Participants) | 12 | 13 | 6 | 14
hour
  Day 1 | 1.04 [0.93 to 5.00] | 1.02 [1.00 to 2.77] | 1.24 [0.97 to 2.17] | 1.05 [0.97 to 3.08]
  Day 8 | 1.21 [0.93 to 3.00] | 1.50 [0.97 to 1.58] | 1.03 [0.95 to 1.42] | 1.13 [0.93 to 5.20]

9. Secondary Outcome: Part A: Volume of Distribution (Vz) for MLN4924
Time Frame: Days 1 and 8: predose and at multiple time-points (up to 72 hours) postdose for Part A
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Part A: MLN4924 8 mg/m^2 + Fluconazole 400 mg | Part A: MLN4924 8 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 15 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 20 mg/m^2 + Itraconazole 200 mg
Number analyzed (Participants) | 12 | 13 | 6 | 14
Liter (L)
  Day 1 | 503 (29.2) | 445 (34.3) | 494 (22.0) | 511 (42.6)
  Day 8: number analyzed (Participants) | 12 | 12 | 6 | 14
  Day 8 | 477 (30.8) | 445 (37.9) | 421 (22.0) | 550 (27.3)

10. Secondary Outcome: Part A: Terminal Phase Elimination Half-life (T1/2) for MLN4924
Time Frame: Days 1 and 8: predose and at multiple time-points (up to 72 hours) postdose for Part A
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Part A: MLN4924 8 mg/m^2 + Fluconazole 400 mg | Part A: MLN4924 8 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 15 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 20 mg/m^2 + Itraconazole 200 mg
Number analyzed (Participants) | 12 | 13 | 6 | 14
hour
  Day 1 | 11.0 (15.7) | 10.6 (20.6) | 9.74 (7.4) | 9.88 (13.8)
  Day 8: number analyzed (Participants) | 12 | 12 | 6 | 14
  Day 8 | 11.6 (14.2) | 13.3 (17.8) | 11.0 (8.0) | 10.7 (9.7)

11. Secondary Outcome: Part A: Blood to Plasma (B/P) Concentration Ratio for MLN4924
Time Frame: Day 1 up to 24 hours post infusion
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part A: MLN4924 8 mg/m^2 + Fluconazole 400 mg | Part A: MLN4924 8 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 15 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 20 mg/m^2 + Itraconazole 200 mg
Number analyzed (Participants) | 12 | 13 | 6 | 13
Ratio
  End of infusion | 51.1 (64.1) | 43.7 (56.9) | 55.2 (30.4) | 35.1 (74.7)
  2 hours post infusion: number analyzed (Participants) | 12 | 13 | 5 | 13
  2 hours post infusion | 69.2 (16.2) | 54.7 (34.7) | 66.5 (30.2) | 48.8 (28.2)
  8 hours post infusion: number analyzed (Participants) | 12 | 13 | 5 | 10
  8 hours post infusion | 71.1 (20.5) | 73.7 (27.5) | 70.7 (38.4) | 56.7 (14.6)
  24 hours post infusion: number analyzed (Participants) | 12 | 13 | 5 | 13
  24 hours post infusion | 71.9 (25.5) | 67.6 (31.3) | 66.3 (17.7) | 58.0 (23.1)

12. Secondary Outcome: Number of Participants Who Experience at Least 1 Treatment-emergent Adverse Event (TEAE) and Serious Adverse Event (SAE)
Time Frame: Baseline up to 30 days after the last dose of study drug (Day 40 for Part A; approximately Cycle 29 for Part B)
Population: The safety population for Part A included all enrolled participants who received at least 1 dose of MLN4924 during Part A and safety population for Part B included all participants who continued to Part B and received at least 1 dose of study drugs during Part B.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: MLN4924 8 mg/m^2 + Fluconazole 400 mg | Part A: MLN4924 8 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 15 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 20 mg/m^2 + Itraconazole 200 mg | Part B: MLN4924 + Docetaxel | Part B: MLN4924 + Carboplatin or Paclitaxel
Number analyzed (Participants) | 13 | 13 | 6 | 19 | 23 | 13
Participants
  TEAE | 13 | 13 | 6 | 18 | 23 | 13
  SAE | 3 | 3 | 2 | 5 | 14 | 6

13. Secondary Outcome: Number of Participants With TEAEs Related to Clinically Significant Laboratory Evaluation Findings
Time Frame: Part A: Baseline up to Day 40; Part B: Baseline up to approximately Cycle 29 Day 35
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: MLN4924 8 mg/m^2 + Fluconazole 400 mg | Part A: MLN4924 8 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 15 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 20 mg/m^2 + Itraconazole 200 mg | Part B: MLN4924 + Docetaxel | Part B: MLN4924 + Carboplatin or Paclitaxel
Number analyzed (Participants) | 13 | 13 | 6 | 19 | 23 | 13
Participants
  Anaemia | 1 | 2 | 0 | 0 | 4 | 2
  Aspartate aminotransferase increased | 0 | 1 | 2 | 0 | 3 | 1
  Alanine aminotransferase increased | 0 | 1 | 1 | 0 | 2 | 1
  Blood creatinine increased | 1 | 0 | 1 | 0 | 0 | 0
  Hyponatraemia | 1 | 0 | 0 | 0 | 0 | 0
  Neutropenia | 0 | 0 | 1 | 0 | 7 | 2
  Hypoalbuminaemia | 1 | 0 | 0 | 0 | 0 | 0
  Leukopenia | 0 | 1 | 0 | 0 | 0 | 0
  Gamma-glutamyltransferase increased | 0 | 1 | 0 | 0 | 0 | 0
  Blood urea increased | 1 | 0 | 0 | 0 | 0 | 0
  Liver function test increased | 0 | 0 | 0 | 1 | 0 | 1
  Neutrophil count decreased | 0 | 0 | 0 | 0 | 2 | 0
  Thrombocytopenia | 0 | 0 | 0 | 0 | 0 | 2
  Platelet count decreased | 0 | 0 | 0 | 0 | 3 | 0
  White blood cell count decreased | 0 | 0 | 0 | 0 | 3 | 1
  Pancytopenia | 0 | 0 | 0 | 0 | 2 | 0
  Hypomagnesaemia | 0 | 0 | 0 | 0 | 0 | 2
  Hyperbilirubinaemia | 0 | 0 | 0 | 0 | 0 | 1
  Lymphocyte count decreased | 0 | 0 | 0 | 0 | 1 | 0
  Blood bilirubin increased | 0 | 0 | 0 | 0 | 0 | 1
  Hypophosphataemia | 0 | 0 | 0 | 0 | 2 | 0
  Hypokalaemia | 0 | 0 | 0 | 0 | 1 | 0
  Hyperuricaemia | 0 | 0 | 0 | 0 | 1 | 0

14. Secondary Outcome: Number of Participants With TEAEs Related to Clinically Significant Vital Sign Findings
Time Frame: Part A: Baseline up to Day 40; Part B: Baseline up to approximately Cycle 29 Day 35
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: MLN4924 8 mg/m^2 + Fluconazole 400 mg | Part A: MLN4924 8 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 15 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 20 mg/m^2 + Itraconazole 200 mg | Part B: MLN4924 + Docetaxel | Part B: MLN4924 + Carboplatin or Paclitaxel
Number analyzed (Participants) | 13 | 13 | 6 | 19 | 23 | 13
Participants
  Tachycardia | 0 | 2 | 0 | 0 | 5 | 3
  Sinus tachycardia | 0 | 0 | 0 | 1 | 0 | 0
  Hypotension | 0 | 0 | 0 | 1 | 7 | 3

15. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Body Weight Measurements
Time Frame: Part A: Baseline up to Day 40; Part B: Baseline up to approximately Cycle 29
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Part A: MLN4924 8 mg/m^2 + Fluconazole 400 mg | Part A: MLN4924 8 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 15 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 20 mg/m^2 + Itraconazole 200 mg | Part B: MLN4924 + Docetaxel | Part B: MLN4924 + Carboplatin or Paclitaxel
Number analyzed (Participants) | 13 | 13 | 6 | 19 | 23 | 13
participants
  Grade 1 AE: 5 < 10% decrease from baseline | 0 | 0 | 0 | 1 | 1 | 1
  Grade 2 AE: 10 - <20% decrease from baseline | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 AE: >=20% decrease from baseline | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Part B: Percentage of Participants With Objective Response
Description: Percentage of participants with objective response based on assessment of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR was defined as complete disappearance of all target lesions. All pathological lymph nodes, both target and non-target, must decrease to normal (short axis less than [<]10 millimeter [mm]). PR was defined as at least 30% decrease under baseline of the sum of diameters of all target lesions.
Time Frame: Baseline up to symptomatic deterioration, progressive disease (PD), treatment discontinuation, or until the study is stopped (approximately Cycle 29)
Population: The response-evaluable population included all participants who received at least 1 dose of study drug in Part B, had measurable disease as entry criteria for Part B, and had at least 1 postbaseline disease assessment. The response-evaluable population where data at specified time points were available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B: MLN4924 + Docetaxel | Part B: MLN4924 + Carboplatin or Paclitaxel
Number analyzed (Participants) | 19 | 9
percentage of participants | 10.5 [1.3 to 33.1] | 22.2 [2.8 to 60.0]

17. Secondary Outcome: Part B: Duration of Response
Description: The duration of response was defined in participants with disease response (CR or PR) as the time between the first documentation of response and progressive disease (PD). Responders without PD will be censored at the last clinical assessment of response. CR was defined as complete disappearance of all target lesions. All pathological lymph nodes, both target and non-target, must decrease to normal (short axis <10 mm). PR was defined as at least 30% decrease under baseline of the sum of diameters of all target lesions. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: Time from the date of first documentation of a response and PD (approximately up Cycle 29)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Part B: MLN4924 + Docetaxel | Part B: MLN4924 + Carboplatin or Paclitaxel
Number analyzed (Participants) | 2 | 2
months | 4.07 (1.440) | 8.46 (1.464)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 30 days after the last dose of study drug (Day 40 for Part A; approximately Cycle 29 for Part B)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Part A: MLN4924 8 mg/m^2 + Fluconazole 400 mg | Part A: MLN4924 8 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 15 mg/m^2 + Itraconazole 200 mg | Part A: MLN4924 20 mg/m^2 + Itraconazole 200 mg | Part B: MLN4924 + Docetaxel | Part B: MLN4924 + Carboplatin or Paclitaxel
All-Cause Mortality (participants affected / at risk) | 2/13 | 3/13 | 1/6 | 2/19 | 6/23 | 1/13
Serious Adverse Events (participants affected / at risk) | 3/13 | 3/13 | 2/6 | 5/19 | 14/23 | 6/13
Other Adverse Events (participants affected / at risk) | 13/13 | 13/13 | 6/6 | 18/19 | 23/23 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: MLN4924 8 mg/m^2 + Fluconazole 400 mg (N=13) | Part A: MLN4924 8 mg/m^2 + Itraconazole 200 mg (N=13) | Part A: MLN4924 15 mg/m^2 + Itraconazole 200 mg (N=6) | Part A: MLN4924 20 mg/m^2 + Itraconazole 200 mg (N=19) | Part B: MLN4924 + Docetaxel (N=23) | Part B: MLN4924 + Carboplatin or Paclitaxel (N=13)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
OESOPHAGEAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
CHOLANGIOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
PANCREATIC CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
METASTATIC SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 0
EMBOLISM (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0
BACTERAEMIA (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
UPPER RESPIRATORY TRACT INFECTIONS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
BLOOD CREATININE INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
VOMITING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
DIAPHRAGMATIC HERNIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
GASTROINTESTINAL PERFORATION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
ASCITES (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
BREAST CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
OESOPHAGEAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
HYPOTENSION (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0
HYPOVOLAEMIC SHOCK (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
CARDIAC ARREST (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
CHEST DISCOMFORT (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
SOFT TISSUE NECROSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
CUSHING'S SYNDROME (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: MLN4924 8 mg/m^2 + Fluconazole 400 mg (N=13) | Part A: MLN4924 8 mg/m^2 + Itraconazole 200 mg (N=13) | Part A: MLN4924 15 mg/m^2 + Itraconazole 200 mg (N=6) | Part A: MLN4924 20 mg/m^2 + Itraconazole 200 mg (N=19) | Part B: MLN4924 + Docetaxel (N=23) | Part B: MLN4924 + Carboplatin or Paclitaxel (N=13)
ANAEMIA (Blood and lymphatic system disorders) | 3 | 3 | 2 | 6 | 5 | 4
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 8 | 2
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
NEUTROPHILIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 2 | 0 | 0 | 4 | 3
SINUS TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
ANGINA PECTORIS (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
PALPITATIONS (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
PHOTOPHOBIA (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
VISION BLURRED (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
EYE ALLERGY (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 3
EYE SWELLING (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
GLAUCOMA (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
LACRIMATION INCREASED (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
OCULAR HYPERAEMIA (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
VISUAL IMPAIRMENT (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
VOMITING (Gastrointestinal disorders) | 3 | 2 | 1 | 6 | 6 | 6
DIARRHOEA (Gastrointestinal disorders) | 0 | 4 | 1 | 6 | 7 | 5
CONSTIPATION (Gastrointestinal disorders) | 3 | 2 | 0 | 3 | 6 | 5
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 3 | 1 | 1 | 1 | 1
NAUSEA (Gastrointestinal disorders) | 3 | 1 | 0 | 2 | 7 | 6
FLATULENCE (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 2 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2 | 0
DYSPEPSIA (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2 | 0
STOMATITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 8 | 3
DYSPHAGIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 0
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
ASCITES (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
CHEILITIS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
DENTAL CARIES (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
ORAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
FATIGUE (General disorders) | 3 | 3 | 1 | 8 | 10 | 5
ASTHENIA (General disorders) | 3 | 2 | 0 | 2 | 5 | 2
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 1 | 0 | 1 | 3 | 2
OEDEMA PERIPHERAL (General disorders) | 0 | 0 | 0 | 3 | 8 | 0
PERIPHERAL SWELLING (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
PYREXIA (General disorders) | 0 | 2 | 0 | 0 | 6 | 2
CATHETER SITE INFLAMMATION (General disorders) | 1 | 0 | 0 | 0 | 1 | 0
GAIT DISTURBANCE (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
ILL-DEFINED DISORDER (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 0 | 0 | 1 | 2 | 0
PAIN (General disorders) | 0 | 0 | 0 | 1 | 3 | 2
CHILLS (General disorders) | 0 | 0 | 0 | 0 | 4 | 0
MALAISE (General disorders) | 0 | 0 | 0 | 0 | 2 | 1
CHEST DISCOMFORT (General disorders) | 0 | 0 | 0 | 0 | 0 | 2
LOCAL SWELLING (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
CATHETER SITE ERYTHEMA (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
CATHETER SITE PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
FACE OEDEMA (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
ANAL INCONTINENCE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
FAECES DISCOLOURED (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
GINGIVAL SWELLING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
MOUTH ULCERATION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
SEASONAL ALLERGY (Immune system disorders) | 0 | 1 | 0 | 1 | 2 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 2 | 0 | 2 | 3 | 2
ORAL HERPES (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
BRONCHITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 2
ORAL CANDIDIASIS (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 0
SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
ABDOMINAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
ANAL ABSCESS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
BREAST CELLULITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
CATHETER SITE ABSCESS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
CELLULITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
FUNGAL SKIN INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
PERINEAL ABSCESS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
SCROTAL ABSCESS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
CATHETER SITE CELLULITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
CONJUNCTIVITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
FOLLICULITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
TINEA PEDIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 2 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 2
PUBIS FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 3 | 0
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
INCISION SITE COMPLICATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
INCISION SITE PAIN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
SKIN WOUND (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
STOMA SITE IRRITATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
BLOOD CREATININE INCREASED (Investigations) | 2 | 0 | 2 | 0 | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 2 | 1 | 0 | 4 | 2
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1 | 2 | 0 | 4 | 2
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 1 | 0 | 1 | 2 | 1
WEIGHT DECREASED (Investigations) | 1 | 0 | 0 | 1 | 2 | 1
AMYLASE DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
BACTERIAL TEST POSITIVE (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
BLOOD SODIUM DECREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
BLOOD UREA INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
BREATH SOUNDS ABNORMAL (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
ELECTROCARDIOGRAM ST SEGMENT DEPRESSION (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
FIBRIN D DIMER INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 | 1 | 0 | 0 | 1 | 1
LIPASE DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
LIVER FUNCTION TEST INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
MICROCOCCUS TEST POSITIVE (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
PANCREATIC ENZYMES DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
WHITE BLOOD CELLS URINE (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 3 | 1
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 2 | 1
PLATELET COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 3 | 0
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
BLOOD CALCIUM DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
BLOOD GLUCOSE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
BLOOD POTASSIUM DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
BLOOD THYROID STIMULATING HORMONE DECREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
ELECTROCARDIOGRAM T WAVE INVERSION (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
THYROXINE DECREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
WEIGHT INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 4 | 3 | 1 | 4 | 10 | 2
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 3 | 2 | 2 | 11 | 3
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 2 | 2 | 3 | 5 | 3
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 | 1 | 1 | 2 | 3 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 | 1 | 0 | 2 | 5 | 0
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 3 | 2
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 5 | 1
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
FLUID RETENTION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
HYPOPHAGIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1 | 4 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 2 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 2
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 2 | 0
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
HAND DEFORMITY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 3
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 3
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 6 | 2
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
JOINT RANGE OF MOTION DECREASED (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
ORAL NEOPLASM BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
TUMOUR ASSOCIATED FEVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 3 | 0 | 0 | 6 | 6 | 3
DIZZINESS (Nervous system disorders) | 1 | 2 | 1 | 4 | 2 | 1
DYSGEUSIA (Nervous system disorders) | 1 | 0 | 0 | 1 | 6 | 1
HYPOAESTHESIA (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 0
APHASIA (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
DISTURBANCE IN ATTENTION (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
SOMNOLENCE (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 | 0 | 0 | 0 | 5 | 3
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 4
AMNESIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
BURNING SENSATION (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
DYSAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
DYSARTHRIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
FACIAL PARALYSIS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
MIGRAINE (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
NEURALGIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
PARAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
SINUS HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
TREMOR (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
ANXIETY (Psychiatric disorders) | 1 | 2 | 0 | 0 | 1 | 2
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 1 | 1 | 0 | 3 | 0
HALLUCINATION (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0
INSOMNIA (Psychiatric disorders) | 2 | 0 | 0 | 0 | 4 | 1
AGITATION (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
IRRITABILITY (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
DEPRESSION (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 1
ABNORMAL DREAMS (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
CHROMATURIA (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
DYSURIA (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0
HAEMATURIA (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
POLLAKIURIA (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1
PROTEINURIA (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
URINARY HESITATION (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 2 | 0
URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 2 | 0
HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
GENITAL RASH (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
VAGINAL LESION (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
VULVOVAGINAL DISCOMFORT (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 3 | 4 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | 1 | 4 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2 | 2
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
PARANASAL SINUS HYPERSECRETION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
PHARYNGEAL ERYTHEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 3 | 1
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1 | 0
BLISTER (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0
ONYCHOMADESIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 3
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0
SKIN LESION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
HYPERTENSION (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0
HAEMATOMA (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
HYPOTENSION (Vascular disorders) | 0 | 0 | 0 | 1 | 6 | 3
LYMPHOEDEMA (Vascular disorders) | 0 | 0 | 1 | 0 | 2 | 0
EMBOLISM (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
FLUSHING (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
ORTHOSTATIC HYPERTENSION (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
EAR PAIN (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
MIDDLE EAR EFFUSION (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
CUSHING'S SYNDROME (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2017-04-12): https://cdn.clinicaltrials.gov/large-docs/70/NCT02122770/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/70/NCT02122770/SAP_001.pdf